CLINICAL TRIAL: NCT02607215
Title: Platinum Retreated in Second- or Third-line Patients With Platinum Sensitive Metastatic Triple Negative Breast Cancer (Randomised, Phase II, NPN Trial)
Brief Title: Platinum Rechallenge in Patients With Platinum-sensitive mTNBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Vice Director of department of medical oncology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2015-19
Record Dates: First submitted 2015-11-16; First posted 2015-11-17 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vinorelbine Plus DDP (Experimental): Vinorelbine:25 mg/m2, D1, D8 every 21 days
  DDP:75 mg/m2, D1 every 21 days
  Interventions: Drug: Vinorelbine; Drug: DDP
- Vinorelbine (Active Comparator): Vinorelbine:30 mg/m2, D1, D8 every 21 days
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine — 25 mg/m2, D1, D8
  Other Names: NVB
Drug: DDP — 75 mg/m2, D1
  Arms: Vinorelbine Plus DDP

SUMMARY:
Platinum Retreated in Patients with Platinum Sensitive mTNBC

DETAILED DESCRIPTION:
Platinum Retreated in Second- or Third-line Patients with Platinum Sensitive Metastatic Triple Negative Breast Cancer (randomised, phase II, NPN trial)

ELIGIBILITY:
Inclusion Criteria:

1. Females with age between 18 and 70 years old
2. Performance status no more than 2
3. Life expectancy longer than 3 months
4. Histological proven unresectable recurrent or advanced breast cancer
5. Triple-negative for estrogen receptor (ER), progestogen receptor (PR), and human epithelial receptor-2 (HER2) by immunohistochemistry (ER <1%, PR <1% and Her2 negative). A negative Her2 gene amplification should be verified by FISH test for those patients with Her2 (2+).
6. Patients must have progressed after 1or 2 prior chemotherapy regimens for metastatic disease, cis/carbo-platin pretreated only 1 previous line prior to randomisation. Platinum sensitive in this study is defined as complete or partial or stable disease following completion (a minimum of 4 treatment cycles) of previous platinum-based chemotherapy and disease progression greater than 3 months after completion of their last dose of platinum chemotherapy (last dose).
7. At least one measurable disease according to the response evaluation criteria in solid tumor (RECIST 1.1)
8. Radiation therapy within 4 weeks prior to enrollment
9. All patients enrolled are required to have adequate hematologic, hepatic, and renal function
10. Be able to understand the study procedures and sign informed consent.

Exclusion Criteria:

1. Patients had prior treatment with vinorelbine
2. Pregnant or lactating women, women of child-bearing potential, unwilling to use adequate contraceptive protection during the process of the study
3. Patients with symptomatic central nervous system metastases are not permitted, except for those with stable and asymptomatic brain metastases who have completed cranial irradiation, and have at least one measurable lesion outside the brain. Radiotherapy should be completed within 4 weeks prior to the registration
4. Treatment with an investigational product within 4 weeks before the first treatment
5. Severe cardiopulmonary insufficiency, severe hepatic and renal dysfunction
6. Uncontrolled serious infection
7. Other active malignancies (including other hematologic malignancies) or other malignancies, except for cured nonmelanoma skin cancer or cervical intraepithelial neoplasia.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2015-11; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 6 weeks

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 weeks
Overall Survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China